CLINICAL TRIAL: NCT02650895
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of CD24Fc When Administered Intravenously in Healthy Adult Subjects
Brief Title: Safety Study of Efprezimod Alfa (CD24Fc, MK-7110) When Administered Intravenously in Healthy Adult Subjects (MK-7110-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oncoimmune, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 7110-001; 1R01NS080821 (NIH); CD24Fc-001 (Other: OncoImmune)
Record Dates: First submitted 2016-01-06; First posted 2016-01-08 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Efprezimod alfa (Experimental): Single dose of efprezimod alfa is administrated as intravenous infusion in one hour. There are 5 dose cohorts, 10mg, 30mg, 60mg, 120mg, 240mg. Each cohort has 6 subjects in efprezimod alfa and 2 subject in placebo.
  Interventions: Biological: Efprezimod alfa
- Saline (Placebo Comparator): Single dose of 100 ml normal saline is administrated as intravenous infusion in one hour.
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: Efprezimod alfa — Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain
  Other Names: CD24IgG; CD24Fc; MK- 7110
  Arms: Efprezimod alfa
Drug: Saline — 0.9% sodium chloride
  Other Names: Normal saline
  Arms: Saline

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single ascending intravenous (IV) doses of efprezimod alfa in healthy adult participants.

DETAILED DESCRIPTION:
This was a Phase I, randomized, double-blind, placebo-controlled, single ascending dose study to assess the safety, tolerability, and pharmacokinetics (PK) of efprezimod alfa in healthy male and female adult participants.

The population for this study was healthy males and females between the ages of 18 and 55 years, inclusive, with a body mass index between 18 kg/m^2 and 30 kg/m^2, inclusive.

A total of 40 participants were enrolled in this study, in 5 cohorts of 8 participants each. Six of the 8 participants in each cohort received study drug and 2 participants received placebo (0.9% sodium chloride, saline). The first cohort was dosed with 10 mg. Succeeding cohorts received 30 mg, 60 mg, 120 mg, and 240 mg of efprezimod alfa or matching placebo and were dosed at least 3 weeks apart to allow for review of safety and tolerability data for each prior cohort. Administration of the next higher dose to a new cohort of participants was permitted only if adequate safety and tolerability had been demonstrated.

In each cohort, the initial 2 participants were 1 study drug recipient and 1 placebo recipient on Day 1 (sentinel participants). Participants 3 to 5 and 6 to 8 were dosed after Day 7 (a minimum of 24 hours apart between the subgroups). Each participant was dosed at least 1 hour apart in the same subgroup. If necessary, dosing of the rest of the participants was delayed pending review of any significant safety issues that may have arisen during the post-dose period involving the first or second subgroups in that cohort. The subsequent cohort was dosed at least 3 weeks after the prior cohort.

The total study duration for each participant, including the screening period, was up to 63 days. Single dose administration occurred on Day 1.

The Screening Visit (Visit 1) occurred up to 21 days prior to the beginning of the active treatment period. After providing informed consent, participants underwent screening procedures for eligibility.

Participants were admitted to the Clinical Pharmacology Unit (CPU) on Day -1 (Visit 2), and the randomized treatment period began on Day 1 following a 10-hour minimum overnight fast. Participants were randomly assigned to treatment with efprezimod alfa or placebo as a single dose. Participants remained confined until the morning of Day 4.

All participants returned to the CPU on Day 7, Day 14, Day 21, Day 28, and Day 42 (±1 day) for follow-up visits (Visit 3, Visit 4, Visit 5, Visit 6, and Visit 7). Visit 7 was the final visit for all participants.

The assessment of safety was based primarily on the frequency of adverse events, clinical laboratory assessments (chemistry, hematology, and urinalysis), physical examinations, vital signs, 12-lead electrocardiograms (ECGs), and continuous telemetry monitoring. The Intent--to--treat (ITT) population was used for all summaries.

PK parameters were calculated using actual collection times. The PK parameters for efprezimod alfa were calculated from the individual serum concentrations profile by noncompartmental approaches.

The PK Evaluable Population was defined as all participants in the ITT Population who had evaluable concentration-time profiles for efprezimod alfa. The PK Evaluable Population was the population used for all PK analyses.

The PK listing, summary, and analysis were performed based on the serum concentration of efprezimod alfa by treatment. Pharmacokinetic parameters were calculated using actual collection times. The PK parameters for efprezimod alfa were calculated from the individual serum concentrations profile by non-compartmental approaches.

The concentration of efprezimod alfa was summarized descriptively at each nominal time point by treatment (e.g., n, mean, standard deviation [SD], coefficient of variation [CV%], standard error, median, minimum, and maximum). Mean concentration (±SD) was plotted on a linear scale against nominal time points by treatment. Geometric mean concentration was plotted on a semi-logarithmic scale against nominal time points. The PK Evaluable Population was used for the summary and individual concentrations.

Individual concentration-time curves for efprezimod alfa were plotted on both a linear and semi-logarithmic scale against actual sampling times by participant.

Pharmacokinetic parameters were summarized for the PK Evaluable Population. All parameters were summarized by treatment with the number of observations, mean, SD, CV%, standard error, median, maximum, and minimum. Geometric mean and geometric CV% were also provided for the summary of area of serum concentration versus time curve (AUC) and maximum serum concentration (Cmax).

Dose proportionality of efprezimod alfa serum PK parameters (AUC and Cmax) was assessed using the power model: y = a Dose β, where y denotes the PK parameter being analyzed and depends on participant. Dose proportionality implies that β = 1 and was assessed by estimated β along with its 90% confidence interval (CI). The exponent, β, in the power model was estimated by regressing the log-transformed PK parameter on log-transformed dose.

The power model was fitted by restricted maximum likelihood using Statistical Analysis System Mixed Model Procedures (SAS Proc Mixed). Both the intercept and slope were fitted as fixed effects. The mean slope was estimated from the power model and the corresponding 90% CI calculated.

The ITT Population consisted of all participants who received at least 1 dose of the study drug. The ITT Population was the primary analysis population for participant information and safety evaluation.

The assessment of safety was based primarily on the frequency and nature of adverse events, clinical laboratory assessments (chemistry, hematology, and urinalysis), physical examinations, vital signs, 12-lead ECGs, and telemetry monitoring. The ITT Population was used for all summaries.

All adverse events were summarized by system organ class, preferred term, and treatment. A list of participants who had serious adverse events (SAEs) and who discontinued from the study due to an adverse event was provided. The number and percentage of participants who experienced at least 1 treatment-emergent adverse event (TEAE) were presented for each system organ class and for each preferred term by treatment. Treatment-emergent adverse events that were considered by the Investigator to be related to study drug were summarized in the same manner. Serious adverse events and adverse events leading to discontinuation from the study were listed separately.

Clinical laboratory evaluations (chemistry, hematology, and urinalysis) were summarized by treatment and visit. Change from baseline was also summarized. Vital signs (blood pressure, heart rate, respiratory rate, and temperature) were summarized by treatment and time point. Change from baseline was also summarized. All physical examination data were listed. Electrocardiogram parameters and the change from baseline were summarized. Overall interpretations were listed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers between the ages of 18 and 55 years, inclusive, in good health based on medical history, physical examination, electrocardiogram (ECG), and routine laboratory tests (blood chemistry, hematology, urinalysis, and drug screen). Any routine laboratory test could be repeated per Investigator judgment;
* Body mass index (BMI) between 18 kg/m2 and 30 kg/m2, inclusive;
* Participants must have been non-smokers or had quit smoking >6 months prior to Screening;
* Women of childbearing potential with a negative urine pregnancy test at Screening who were not breastfeeding, did not plan to become pregnant during the study, and agreed to use dual methods of birth control during the study (i.e., 2 of the following: diaphragm or cervical cap with spermicide, intrauterine device [IUD] hormonal contraceptives [stable for at least 3 months prior to Screening], male partner using condom with spermicide) from Day 1 until 60 days following the administration of study drug; or female participants of non-childbearing potential were either surgically sterile (hysterectomy, bilateral oophorectomy, or bilateral tubal ligation) or >1 year post-menopausal with a follicle-stimulating hormone (FSH) in the post menopausal range (post-menopausal taking hormone replacement therapy [stable for at least 3 months prior to Screening] did not require an FSH level);
* All male participants were required to use barrier contraception (condom with spermicide) in addition to having their female partner (if of childbearing potential) use another acceptable form of contraception (IUD, diaphragm with spermicide, hormonal contraceptives [stable for at least 3 months prior to Screening]) from Day 1 until 60 days following the last administration of study drug;
* Negative alcohol, cotinine, and drug screen;
* Willing to abstain from alcohol for 48 hours prior to any visit;
* Willing and able to be confined to the CPU as required by the protocol;
* Willing and able to comply with the investigational nature of the study and able to communicate well with the Principal Investigator and clinical staff; and
* Ability to comprehend and willingness to provide written informed consent in accordance with institutional and regulatory guidelines.

Exclusion Criteria:

* Participants with evidence or history of clinically significant immunologic, hematologic, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies), surgical conditions, cancer or any other condition that, in the Investigator's opinion, might significantly interfere with the absorption, distribution, metabolism, or excretion of the study drug;
* Participants who had received any investigational drug or device within 30 days or less than 5 half-lives of investigational drug prior to dosing;
* Participants taking any prescription or over-the-counter medications within 7 days prior to dosing, or were not willing to refrain from these medications throughout the study period;
* Participants who had a history of alcoholism or drug abuse within 2 years prior to dosing;
* Participants with a typical consumption of 14 alcoholic drinks weekly;
* Participants who had a history of or positive tests for human immunodeficiency virus (HIV) or hepatitis C virus (HCV), or participants who had a positive hepatitis B surface antigen (HBsAg) at Screening;
* Participants who had donated blood or blood products within 30 days prior to dosing;
* Participants with inadequate venous access;
* Participants with an aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 the upper limit of normal (ULN) at Screening or Day -1;
* Participants with a total bilirubin >1.5 ULN at Screening or Day -1;
* Participants who were currently undergoing treatment with weight loss medication or prior weight loss surgery (e.g., gastric bypass surgery);
* Participants who had poor mental function or any other reason to expect participant difficulty in complying with the requirements of the study; or
* Participants who had a history or presence of any medical condition or disease that, in the opinion of the Investigator, could interfere with the conduct of the study or would put the participant at unacceptable risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-06-02 (Actual); Primary Completion 2015-01-15 (Actual); Study Completion 2015-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Medpace Clinical Pharmacology Unit (CPU), Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Wang X, Liu M, Zhang J, Brown NK, Zhang P, Zhang Y, Liu H, Du X, Wu W, Devenport M, Tao W, Mao-Draayer Y, Chen GY, Chen YE, Zheng P, Liu Y. CD24-Siglec axis is an innate immune checkpoint against metaflammation and metabolic disorder. Cell Metab. 2022 Aug 2;34(8):1088-1103.e6. doi: 10.1016/j.cmet.2022.07.005. PMID 35921817
- See also: Description: Merck Oncology Clinical Trials Information — http://merckoncologyclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study Period: 32 weeks. Initiation Date: 02 June 2014. Completion Date: 15 January 2015. Study site: Clinical Pharmacology Unit, Medpace Inc. Cincinnati, Ohio.
Pre-assignment Details: Diagnosis and Main Criteria for Inclusion: The population for this study was healthy males and females between the ages of 18 and 55 years, inclusive, in good health based on medical history, physical examination, electrocardiogram (ECG), and routine laboratory tests, with a body mass index between 18 kg/m2 and 30 kg/m2, inclusive.
Groups:
- Saline: Single dose of 100 ml normal saline is administrated as intravenous infusion in one hour. Saline: 0.9% sodium chloride
- CD24Fc 10 mg: Single dose of 10 mg CD24Fc diluted in 0.9% sodium chloride in final volume of 100 ml is administrated as intravenous infusion in one hour. CD24Fc: Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain.
- CD24Fc 30 mg: Single dose of 30 mg CD24Fc diluted in 0.9% sodium chloride in final volume of 100 ml is administrated as intravenous infusion in one hour. CD24Fc: Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain.
- CD24Fc 60 mg: Single dose of 60 mg CD24Fc diluted in 0.9% sodium chloride in final volume of 100 ml is administrated as intravenous infusion in one hour. CD24Fc: Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain.
- CD24Fc 120 mg: Single dose of 120 mg CD24Fc diluted in 0.9% sodium chloride in final volume of 100 ml is administrated as intravenous infusion in one hour. CD24Fc: Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain.
- CD24Fc 240 mg: Single dose of 240 mg CD24Fc diluted in 0.9% sodium chloride in final volume of 100 ml is administrated as intravenous infusion in one hour. CD24Fc: Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain.
Period: Overall Study
Arm/Group | Saline | CD24Fc 10 mg | CD24Fc 30 mg | CD24Fc 60 mg | CD24Fc 120 mg | CD24Fc 240 mg
Started | 10 | 6 | 6 | 6 | 6 | 6
Completed | 10 | 5 | 6 | 6 | 6 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saline | CD24Fc 10 mg | CD24Fc 30 mg | CD24Fc 60 mg | CD24Fc 120 mg | CD24Fc 240 mg | Total
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (9.87) | 33.2 (6.65) | 30.0 (11.37) | 33.5 (7.71) | 43.3 (9.40) | 35.5 (7.77) | 34.8 (9.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 3 | 4 | 2 | 1 | 17
  Male | 7 | 2 | 3 | 2 | 4 | 5 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 10 | 6 | 6 | 5 | 6 | 5 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 4 | 5 | 4 | 5 | 3 | 28
  White | 3 | 2 | 1 | 1 | 1 | 2 | 10
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 6 | 6 | 6 | 6 | 6 | 40

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Safety Based Primarily on the Frequency and Nature of Adverse Events, Clinical Laboratory Assessments (Chemistry, Hematology, and Urinalysis), Physical Examinations, Vital Signs, 12-lead Electrocardiograms (ECGs), and Telemetry Monitoring
Description: List of adverse events in the form of frequency and grade. Assessment of safety based primarily on the frequency and nature of adverse events, clinical laboratory assessments (chemistry, hematology, and urinalysis), physical examinations, vital signs, 12-lead ECGs, and telemetry monitoring from pre-dosing to day 42 visits. The data include all treatment-emergent adverse events (TEAEs) including specific drug-related TEAEs.
Time Frame: Up to 42 days after treatment
Population: The analysis population included all participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Saline | CD24Fc 10 mg | CD24Fc 30 mg | CD24Fc 60 mg | CD24Fc 120 mg | CD24Fc 240 mg
Number analyzed (Participants) | 10 | 6 | 6 | 6 | 6 | 6
Participants
  Subjects without any drug-related TEAE | 9 | 4 | 5 | 5 | 6 | 6
  Nervous system disorders: Headache | 1 | 2 | 1 | 0 | 0 | 0
  Cardiac disorders: Ventricular tachycardia | 0 | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Serum Concentration of CD24Fc Over Time
Description: Measurement of serum CD24Fc concentration at different time points after administration.
Time Frame: Up to 42 days after treatment
Population: The analysis population included all participants who received at least one dose of study medication and who had evaluable concentration data for CD24Fc.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | CD24Fc 10 mg | CD24Fc 30 mg | CD24Fc 60 mg | CD24Fc 120 mg | CD24Fc 240 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/ml
  Pre-dose | 12.8 (31.36) | 9.2 (22.49) | 25.7 (44.48) | 0.0 (0.00) | 0.0 (0.00)
  1 hour post-dose | 2464.7 (571.94) | 9715.9 (1716.63) | 30082.5 (7178.61) | 49491.7 (8113.51) | 94091.3 (13576.66)
  2 hours post-dose | 2245.3 (527.14) | 8566.7 (1037.74) | 25178.0 (6339.22) | 49598.0 (11087.03) | 87735.2 (13424.35)
  12 hours post-dose: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6
  12 hours post-dose | 1680.6 (191.57) | 5842.6 (612.76) | 17068.8 (4353.50) | 26906.5 (7418.39) | 55358.3 (10202.10)
  24 hours post-dose: number analyzed (Participants) | 6 | 6 | 5 | 6 | 6
  24 hours post-dose | 1506.0 (279.92) | 5251.0 (449.67) | 14109.8 (4335.70) | 25874.5 (7187.38) | 46554.7 (7213.90)
  72 hours post-dose | 996.1 (259.34) | 3615.6 (538.01) | 9792.5 (1186.99) | 15552.3 (4930.29) | 31793.7 (4360.83)
  Day 7: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Day 7 | 754.4 (183.84) | 1941.5 (138.83) | 6585.3 (2861.77) | 11649.3 (4299.71) | 21963.5 (3042.93)
  Day 14: number analyzed (Participants) | 5 | 6 | 6 | 6 | 5
  Day 14 | 419.5 (112.20) | 1261.8 (108.92) | 2712.6 (762.02) | 7336.7 (2552.98) | 13083.8 (2081.62)
  Day 28: number analyzed (Participants) | 5 | 6 | 6 | 6 | 6
  Day 28 | 218.5 (69.86) | 672.3 (80.26) | 1199.6 (298.24) | 2969.4 (1251.53) | 6162.3 (909.27)
  Day 42 | 87.3 (35.07) | 315.0 (73.96) | 643.5 (244.95) | 1563.8 (641.24) | 2799.3 (463.22)

3. Secondary Outcome: Maximum Serum Concentration (Cmax) of CD24Fc
Description: Assessment of CD24Fc pharmacokinetics based on serum CD24Fc concentration at different time points after administration to determine drug Cmax. Cmax was defined as the maximum concentration of CD24Fc observed in serum following administration of CD24Fc.
Time Frame: Up to 42 days after treatment
Population: The analysis population included all participants who received at least one dose of study medication and who had evaluable pharmacokinetic Cmax data for CD24Fc.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | CD24Fc 10 mg | CD24Fc 30 mg | CD24Fc 60 mg | CD24Fc 120 mg | CD24Fc 240 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng/mL | 2495 (576) | 9735 (1715) | 30083 (7179) | 52435 (9910) | 95865 (10734)

4. Secondary Outcome: Area Under the Serum Concentration Curve From 0-42 Days (AUC 0-42d) of CD24Fc
Description: AUC was defined as the area of serum concentration versus time curve from time zero to 42 days (AUC 0-42d). Assessment of AUC 0-42d was based on CD24Fc concentration measured at different time points after administration of CD24Fc.
Time Frame: Up to 42 days after treatment
Population: The analysis population included all participants who received at least one dose of study medication and who had evaluable pharmacokinetic AUC 0-42d data for CD24Fc.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | CD24Fc 10 mg | CD24Fc 30 mg | CD24Fc 60 mg | CD24Fc 120 mg | CD24Fc 240 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 423061 (99615) | 1282430 (88798) | 3226255 (702862) | 6541501 (2190944) | 12704705 (1918596)

5. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of CD24Fc
Description: t1/2 was defined as the time required to divide the serum concentration by two after reaching maximum concentration (Cmax), following administration of CD24Fc.
Time Frame: Up to 42 days after treatment
Population: The analysis population included all participants who received at least one dose of study medication and who had evaluable t1/2 data for CD24Fc.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | CD24Fc 10 mg | CD24Fc 30 mg | CD24Fc 60 mg | CD24Fc 120 mg | CD24Fc 240 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
hr | 280.83 (22.37) | 327.10 (41.32) | 279.82 (65.59) | 286.45 (23.38) | 285.33 (24.33)

ADVERSE EVENTS:
Time Frame: Up to 42 days after treatment
Description: The analysis population included all participants who received at least one dose of study medication.
Groups:
- CD24Fc 10 mg: Single dose of 10 mg CD24Fc is administrated as intravenous infusion in one hour. CD24Fc: Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain
- CD24Fc 30 mg: Single dose of 30 mg CD24Fc is administrated as intravenous infusion in one hour. CD24Fc: Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain
- CD24Fc 60 mg: Single dose of 60 mg CD24Fc is administrated as intravenous infusion in one hour. CD24Fc: Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain
- CD24Fc 120 mg: Single dose of 120 mg CD24Fc is administrated as intravenous infusion in one hour. CD24Fc: Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain
- CD24Fc 240 mg: Single dose of 240 mg CD24Fc is administrated as intravenous infusion in one hour. CD24Fc: Recombinant fusion protein consisting of the extracellular domain of mature human CD24 linked to the human immunoglobulin G1 (IgG1) Fc domain
Arm/Group | Saline | CD24Fc 10 mg | CD24Fc 30 mg | CD24Fc 60 mg | CD24Fc 120 mg | CD24Fc 240 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/6 | 0/6 | 1/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 6/10 | 2/6 | 3/6 | 2/6 | 3/6 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline (N=10) | CD24Fc 10 mg (N=6) | CD24Fc 30 mg (N=6) | CD24Fc 60 mg (N=6) | CD24Fc 120 mg (N=6) | CD24Fc 240 mg (N=6)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Saline (N=10) | CD24Fc 10 mg (N=6) | CD24Fc 30 mg (N=6) | CD24Fc 60 mg (N=6) | CD24Fc 120 mg (N=6) | CD24Fc 240 mg (N=6)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory tract infections (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No